CLINICAL TRIAL: NCT05723640
Title: Phase I, Open-Label Study of the Safety and Dosimetry of a 4-Dose Regimen of Escalating Doses of 177Lu-LNC1004 Injection in Adult Patients With Advanced Fibroblast Activation Protein (FAP)-Positive Solid Tumors
Brief Title: The Safety and Dosimetry Study of 177Lu-LNC1004 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yantai LNC Biotechnology Singapore PTE. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-LNC1004-001
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor, Unspecified, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 177Lu-LNC1004 Injection group 1 (Experimental): 177Lu-LNC1004 Injection, a single dose of 30mCi will be administered every 6 weeks, for a total of 2 cycles.
  Interventions: Drug: 177Lu-LNC1004 Injection group 1 radionuclide therapy
- 177Lu-LNC1004 Injection group 2 (Experimental): 177Lu-LNC1004 Injection, a single dose of 60mCi will be administered every 6 weeks, for a total of 2 cycles.
  Interventions: Drug: 177Lu-LNC1004 Injection group 2 radionuclide therapy
- 177Lu-LNC1004 Injection group 3 (Experimental): 177Lu-LNC1004 Injection, a single dose of 80mCi will be administered every 6 weeks, for a total of 2 cycles.
  Interventions: Drug: 177Lu-LNC1004 Injection group 3 radionuclide therapy
- 177Lu-LNC1004 Injection group 4 (Experimental): 177Lu-LNC1004 Injection, a single dose of 100mCi will be administered every 6 weeks, for a total of 2 cycles.
  Interventions: Drug: 177Lu-LNC1004 Injection group 4 radionuclide therapy

INTERVENTIONS:
Drug: 177Lu-LNC1004 Injection group 1 radionuclide therapy — The treatment regimen will consist of a single dose 30mCi intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles, the dose per cycle will be fixed.
  Arms: 177Lu-LNC1004 Injection group 1
Drug: 177Lu-LNC1004 Injection group 2 radionuclide therapy — The treatment regimen will consist of a single dose 60mCi intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles, the dose per cycle will be fixed.
  Arms: 177Lu-LNC1004 Injection group 2
Drug: 177Lu-LNC1004 Injection group 3 radionuclide therapy — The treatment regimen will consist of a single dose 80mCi intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles, the dose per cycle will be fixed.
  Arms: 177Lu-LNC1004 Injection group 3
Drug: 177Lu-LNC1004 Injection group 4 radionuclide therapy — The treatment regimen will consist of a single dose 100mCi intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles, the dose per cycle will be fixed.
  Arms: 177Lu-LNC1004 Injection group 4

SUMMARY:
This proposal is a phase I, open-label study of a 4-Dose Regimen of Escalating Doses of 177Lu-LNC1004 Injection in patients with recurrent or metastatic, fibroblast activation protein-positive solid tumors.

In the clinical development, we aim to demonstrate the following:

* 177Lu-LNC1004 Injection is safe and tolerable at therapeutic dose.
* Determination of dose(s) to be used in the expansion phase. The treatment regimen will consist of a single dose intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles. The dose per cycle will be fixed for each patient and will be escalated in 4 different dose levels

DETAILED DESCRIPTION:
This proposal is a phase I, open-label study of a 4-Dose Regimen of Escalating Doses of 177Lu-LNC1004 Injection in patients with recurrent or metastatic, fibroblast activation protein-positive solid tumors. The treatment regimen will consist of a single dose intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles. The dose per cycle will be fixed for each patient and will be escalated in 4 different dose levels, from 30 mCi to 100 mCi (1.11 - 3.7 GBq).

This classic 3+3 design includes 3 patients for the first dose level group. If no DLT occurs, 3 patients will be enrolled at the next dose level. If a DLT occurs at a certain dose level, 3 additional patients will be enrolled at the previous dose level. The highest dose with no more than 1 DLT out of 6 patients will be defined as MTD. If there is no MTD observed after the dose escalation up to 100 mCi, a comprehensive evaluation should be made by investigator and sponsor to determine whether an escalation to a higher dose can be conducted or not based on the known safety, radiation dose and efficacy characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and sign an approved informed consent form (ICF).
* Patients must have the ability to understand and comply with all protocol requirements.
* Aged 21 years or older
* Patients must have histological, pathological, and/or cytological confirmation of advanced/metastatic solid tumor that is refractory to or has progressed following prior treatment and based on the current guidelines, there is no recommended treatment
* Measurable disease as defined by Response Criteria in Solid Tumors (RECIST) version 1.1
* Overexpression of fibroblast activation protein of the target lesions at 68Ga-FAPI-46 positron emission tomography (PET)/computed tomography (CT) with positive uptake (higher than adjacent background).
* Eastern Cooperative Oncology Group (ECOG) performance status (ECOG PS) score of 0 or 1
* Adequate organ function as defined by:

  1. Creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula)
  2. Hemoglobin (Hb) > 9.0g/dL
  3. Absolute neutrophil count (ANC) > 1.5 x 10^9/L
  4. Platelets ≥100 x 109/L
  5. International normalized ratio (INR) < 1.5 for patients that are not on warfarin
  6. Prothrombin time (PTT) < 2 x ULN
  7. Total bilirubin < 1.5 x ULN
  8. Serum albumin > 2.8 g/dL
  9. Alanine aminotransferase (ALT) <3 x ULN, or <5 x ULN if deemed related to liver metastases from solid tumor
  10. Aspartate aminotransferase (AST) <3 x ULN, or <5 x ULN if deemed related to liver metastases from solid tumor
* All other toxicity parameters must be NCI-CTCAE v.5.0 Grade 0 or 1
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at study entry. Subjects not considered WOCBP are those without menses for ≥ 12 consecutive months, and those who have undergone hysterectomy and/or bilateral salpingo-oophorectomy. WOCBP must be willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study and 6 months after the last dose of treatment.
* Male participants with partners of childbearing potential are required to use barrier contraception in addition to having their partner use another method of contraception during the study and for 6 months after the last dose of treatment. Male participants will also be advised to abstain from sexual intercourse with pregnant or lactating women, or to use condoms.
* Previous surgery no less than 4 weeks prior to study entry.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-LNC1004 as assessed from medical records
* Participant has had prior chemotherapy or radical radiotherapy within 4 weeks before the first administration of study drug
* Participant has had prior targeted cancer therapy, immunotherapy, or treatment with an investigational anticancer agent ≤ 14 days prior to receiving study treatment (≤ 28 days prior in case of checkpoint inhibitor or other antibody therapies) before the first administration of study drug.
* Received prior radiopharmaceutical therapy or radioembolization, or prior extensive external beam radiation therapy (EBRT) to bone marrow or any prior EBRT to kidney, or received any EBRT within 2 weeks prior to administration of study treatment
* Participant has not fully recovered from major surgery or significant traumatic injury prior the first dose of study drug or expects to have major surgery during the study period or within 3 months after the last dose of study drug.
* Life expectancy < 6 months as assessed by the treating physician
* > 80% liver involvement by tumor
* > 25% bone marrow involvement by tumor
* Clinically significant abnormalities on electrocardiogram (ECG) at screening including QTcF > 470 ms regardless of sex or subjects who cannot tolerate high volume load.
* Toxicities from prior therapies that have not resolved to grade 1 or grade 0
* Active and clinically significant bacterial, fungal, or viral infection, including hepatitis B (HBV), hepatitis C (HBC), know human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
* Known brain metastases and/or carcinomatous meningitis, unless these metastases have been treated and stabilized
* Uncontrolled diabetes mellitus as defined by a HbA1c >9%
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior external beam radiation therapy involving >25% of the bone marrow
* Unmanageable urinary incontinence rendering the administration of 177Lu-LNC1004 unsafe
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and with no evidence of recurrence
* Unable to comply with relevant contact precautions post 177Lu-LNC1004 treatment
* Any other condition that may increase the risk associated with study participation or interfere with its interpretation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
the safety of 177Lu-LNC1004 Injection | through study completion, assessed up to 2 years.
  To evaluate the safety of 177Lu-LNC1004 Injection assessed from the number of patients with treatment-related adverse events using CTCAE v5.0.
To identify the dose-limiting toxicities (DLTs) | through cycle 1, an average of 6 weeks
  To identify the dose-limiting toxicities (DLTs) of escalating doses of 177Lu-LNC1004 up to 100 mCi (3.7 GBq) administered intravenously to patients in the first cycle.
To determine if the MTD is among the explored dose levels and identify the expansion phase dose | through study completion, assessed up to 2 years.
  To determine if the maximum tolerated dose is among the explored dose levels and identify the expansion phase dose of 177Lu-LNC1004 Injection.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Cancer Institute, Singapore National University Hospital, Singapore., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No